CLINICAL TRIAL: NCT06383806
Title: Imagery Rehearsal Therapy for the Treatment of Nightmares in Narcolepsy: A Pilot Randomized Controlled Trial
Brief Title: Decreasing Nightmares in Adults With Narcolepsy
Acronym: DAWN
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Utah (Other)
Responsible Party: Principal Investigator, Jennifer Mundt, Assistant Professor, University of Utah
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: IRB_00188162; 372-SR-25 (Other Grant/Funding Number: American Academy of Sleep Medicine Foundation)
Record Dates: First submitted 2024-04-22; First posted 2024-04-25 (Actual); Last update posted 2025-07-15 (Actual); Status verified 2025-07

CONDITIONS: Narcolepsy; Narcolepsy Type 1; Narcolepsy With Cataplexy; Narcolepsy Without Cataplexy; Nightmare; Nightmare Disorder With Associated Other Sleep Disorder
Keywords: Imagery Rehearsal Therapy; Cognitive Behavioral Therapy for Nightmares
MeSH Terms: conditions — Narcolepsy | interventions — Cognitive Behavioral Therapy

STUDY DESIGN:
Intervention Model Description: Waitlist control
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Treatment (Experimental): The Treatment arm will receive the intervention immediately following the first assessment.
  Interventions: Behavioral: Imagery Rehearsal Therapy (IRT)
- Waitlist (Other): The Waitlist arm will undergo a waiting period following the first assessment and then will receive the treatment after the second assessment.
  Interventions: Behavioral: Imagery Rehearsal Therapy (IRT)

INTERVENTIONS:
Behavioral: Imagery Rehearsal Therapy (IRT) — The intervention will consist of 7 therapy sessions (once per week for 7 weeks) which will be delivered via videoconference. During the sessions, participants will learn techniques for managing and changing nightmares.
  Other Names: Cognitive Behavioral Therapy for Nightmares (CBT-N)

SUMMARY:
The purpose of this clinical trial is learn whether a behavioral (non-medication) treatment can reduce nightmares in adults with narcolepsy. All participants will receive the treatment and will complete three assessments. Half of the participants will receive the treatment after the first assessment, and half will receive it after the second assessment. Romantic partners of participants with narcolepsy will also be eligible to enroll in the study. Partners will complete three assessments but will not participate in the treatment.

ELIGIBILITY:
PARTICIPANTS WITH NARCOLEPSY/NIGHTMARES

Inclusion Criteria:

* Diagnosis of narcolepsy type 1 or narcolepsy type 2
* Nightmare frequency of ≥1 times per week
* Age 18 or older
* Able to speak, read, and write in English
* Live in the United States
* Sleep and psychiatric medications stable for ≥ 1 month and willing to keep medications stable for the duration of the study

Exclusion Criteria:

* Currently engaged in trauma- or sleep-related psychotherapy
* Previous behavioral treatment for nightmares
* Medical, psychiatric, or cognitive condition which would interfere with ability to engage in the treatment
* Untreated moderate-severe sleep apnea

PARTICIPANTS WHO ARE PARTNERS OF SOMEONE WITH NARCOLEPSY

Inclusion Criteria:

* Live with a romantic partner who meets the above criteria and has agreed to participate in the study
* Age 18 or older
* Able to speak, read, and write in English
* Live in the United States

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2025-06-06 (Actual); Primary Completion 2027-09 (Estimated); Study Completion 2027-09 (Estimated)

PRIMARY OUTCOMES:
Disturbing Dream and Nightmare Severity Index (DDNSI) | Completed at each of the three assessments (baseline, 10 weeks, 19 weeks)
  The DDNSI is a questionnaire which measures the severity of nightmares.
Nightmare frequency (sleep diary) | Completed at each of the three assessments (baseline, 10 weeks, 19 weeks)
  The number of nightmares experienced each day will be collected on daily sleep diaries completed during each assessment period.

SECONDARY OUTCOMES:
PROMIS Anxiety | Completed at each of the three assessments (baseline, 10 weeks, 19 weeks)
  Questionnaire which measures the severity of anxiety symptoms.
PROMIS Depression | Completed at each of the three assessments (baseline, 10 weeks, 19 weeks)
  Questionnaire which measures the severity of depressive symptoms.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Utah, Salt Lake City, Utah, United States

IPD SHARING:
Plan to Share IPD: No